CLINICAL TRIAL: NCT03646370
Title: Assessing Virologic Success and Metabolic Changes in Patients Switching From a TDF to TAF Containing Antiretroviral Therapy Regimen
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 18G.433
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: HIV-1-infection; Metabolic Syndrome; Cardiovascular Diseases; Weight Gain; Renal Function Abnormal; Hyperglycemia
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Weight Gain; Hyperglycemia | interventions — tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Patients with HIV infection who are virally suppressed receiving a tenofovir disoproxil fumarate-based antiretroviral therapy regimen that switched to tenofovir alafenamide without switching any other components of their treatment regimen.

SUMMARY:
Switching patients with HIV infection from tenofovir disoproxil fumarate (TDF) to a tenofovir alafenamide (TAF) based drug regimen can provide many safety benefits including preserving bone mineral density and kidney function. This study will examine metabolic changes that patients may encounter due to the switch in medication regimens and the maintenance of viral suppression.

DETAILED DESCRIPTION:
Many providers of HIV medicine are switching patients from TDF to TAF containing ART regimens for safety reasons including significant improvements in bone health and kidney function that have been demonstrated in clinical trials.1-3 Multiple studies have evaluated the efficacy and safety of switching from TDF to TAF based regimens, but most allowed other components of the ART regimen to change in addition to TDF which may confound study results. For example, a recent meta-analysis demonstrated that TDF accompanied by ritonavir or cobicistat boosting was associated with higher risks of bone and renal adverse events and lower rates of virologic suppression in comparison to TAF. In contrast, when ritonavir and cobicistat were not used, there were not efficacy differences and only marginal safety differences between tenofovir agents.4 Additionally, measures of treatment success aside from maintaining virologic suppression including requirements for additional regimen changes due to tolerability, cost and access have not been formally evaluated. Furthermore, aside from renal function and bone health, comprehensive evaluations of metabolic changes following TDF to TAF switches have not been performed. Specifically, alterations in weight, body mass index, and glycemic control have not been studied in patients switching from TDF to TAF in clinical trials and changes in cholesterol and cardiovascular disease risk have had only minimal assessment.5 Weight gain most commonly occurs following the initiation of ART in treatment naïve patients, but has been noted in virologically suppressed patients making certain ART changes. Weight gain following TDF to TAF switches was not measured in clinical trials, but has been noted anecdotally within our clinic population and is believed to warrant additional investigation.

In terms of cholesterol and cardiovascular disease risk, previous clinical trials have identified differences in serum cholesterol measurements in patients receiving TDF and TAF, but formal assessments of the resulting potential differences in cardiovascular disease risk have not occurred:

* The first trial was a phase II, randomized, double-blind, double-dummy, multi-center study that compared the safety and efficacy of TAF and TDF.6 The active-controlled arm received elvitegravir 150mg, cobicistat 150mg, emtricitabine 200mg, and TDF 200mg (E/C/F/TDF). The study arm received elvitegravir, cobicistat, emtricitabine, and TAF (E/C/F/TAF). Subjects receiving E/C/F/TAF experienced more Grade 3 or 4 increases in low-density lipoprotein cholesterol (LDL) (9% vs. 3%). However, the median increase in fasting LDL was similar between groups (+17 vs. +11 mg/dL, p=0.11). Significant differences were observed for total cholesterol (+30 vs +17 mg/dL, p=0.007) and high-density lipoprotein (HDL) (+7 vs +3 mg/dL, p=0.023), but the total cholesterol:HDL ratio remained similar for both treatment arms.
* A second phase II, randomized, double-blind, double-dummy multicenter trial compared darunavir 800mg/cobicistat 150mg/emtricitabine 200mg/TAF 10mg (D/C/F/TAF) to darunavir 800mg, cobicistat 150mg, and co-formulated emtricitabine 200mg/TDF 300mg (D+C+F/TDF).7 More than 230 subjects were screened, and 153 were randomized 2:1 to receive either D/C/F/TAF (n=103) or D+C+F/TDF (n=50). The primary efficacy outcome was virologic suppression at weeks 24 and 48. Safety and tolerability were assessed through renal, bone, and metabolic measurements. At the end of the trial, fasting lipid changes from baseline were greater in the TAF group at week 48 for total cholesterol (+40 vs. +5 mg/dL, p<0.001), LDL (+26 vs. +4 mg/dL, p<0.001), HDL (+7 vs. +3 mg/dL, p=0.009), and triglycerides (+29 vs. -5 mg/dL, p=0.007). The total change in total cholesterol:HDL ratio was again comparable between groups (0 vs. -0.2, p=0.15).
* A randomized, active-controlled, open-label study assessed the safety and efficacy of switching virologically suppressed HIV-infected patients from their TDF-based regimen to E/C/F/TAF.8 The study assessed 601 patients who were randomized 2:1 to receiving E/C/F/TAF (n=402) or maintain their current regimen of FTC/TDF plus atazanavir boosted with cobicistat or ritonavir (n=199). Again, patients receiving E/C/F/TAF had statistically significant median increases in total cholesterol (+23 vs. + 5 mg/dL, p<0.001) and in LDL (+9 vs -1 mg/dL, p<0.001). Additionally, the proportion of patients who initiated lipid-modifying agents was greater in the E/C/F/TAF group but was not statistically significant (8.5% vs. 5%, p=0.14).

In each trial, it is evident that patients receiving TAF have greater elevations in serum cholesterol levels in comparison to TDF. However, the majority of trials also note that the total cholesterol:HDL ratio appears to be similar among TDF and TAF recipients. This value has been used by investigators to suggest that differences in cardiovascular disease risk are unlikely to be present among TDF and TAF recipients despite considerable increases in total cholesterol, LDL and triglycerides levels in TAF recipients. The current ACC/AHA guidelines on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults, do not recommend the use of the total cholesterol:HDL ratio to determine risk for cardiovascular disease.9 Rather, they recommend using the atherosclerotic cardiovascular disease (ASCVD) scoring system, which incorporates cholesterol values in additional to other factors that influence cardiovascular disease risk. This level of cardiovascular disease risk assessment has not been performed and assessed for TAF and TDF in clinical trials.

The current study is significant because it will add to the current clinical knowledge of TAF in terms of efficacy, safety and tolerability. It will evaluate treatment success when patients have isolated TDF to TAF switches by analyzing virologic and immunologic responses in addition to the need for subsequent regimen changes due to poor tolerability, cost restriction or access limitations. This study will also provide a comprehensive assessment of potential metabolic changes following isolated TDF to TAF changes. This includes changes in the incidence of metabolic syndrome, alterations in cholesterol and cardiovascular disease risk, changes in weight and body mass index (BMI), and changes in glycemic control and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV who are virally suppressed receiving a tenofovir disoproxil fumarate-based antiretroviral therapy regimen that switched to tenofovir alafenamide without switching any other components of their medications.

Exclusion Criteria:

* Patients are excluded if their switch was prior to 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV infection who are on antiretroviral therapy and virally suppressed who have switched one medication within their treatment regimen for safety reasons.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Changes in weight | 1 year
  Changes in weight will be determined through comparisons of average baseline and endpoint weights
Changes in metabolic syndrome | 1 year
  Changes in the presence of metabolic syndrome will be determined through comparisons of baseline and endpoint modified metabolic syndrome diagnostic criteria defined by the American Heart Association.
Changes in glycemic control | 1 year
  Changes in glycemic control will be determined through comparisons of baseline and endpoint fasting blood glucose and hemoglobin A1C levels
Changes in kidney function | 1 year
  Changes in kidney function will be determined through comparisons of baseline and endpoint creatinine clearance estimations.
Changes in cholesterol | 1 year
  Changes in cholesterol will be determined through comparisons of baseline and endpoint total cholesterol levels.
Changes in 10-year cardiovascular disease risk | 1 year
  Each patient's estimated 10-year cardiovascular disease risk will be calculated at baseline and endpoint after the ART regimen switch using the ASCVD scoring system.

SECONDARY OUTCOMES:
Treatment success | 1 year
  * Patients will meet criteria for treatment success after their ART regimen switch if they maintain viral suppression and adherence to their TAF regimen for 12 months without having to incur additional ART switches due to toxicity, poor tolerability, cost restriction or access limitations.
  * Subgroup analyses will be performed to investigate factors associated with a lack of treatment success, if present, including the presence of a boosting agent within the ART regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jeffeson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills A, Arribas JR, Andrade-Villanueva J, DiPerri G, Van Lunzen J, Koenig E, Elion R, Cavassini M, Madruga JV, Brunetta J, Shamblaw D, DeJesus E, Orkin C, Wohl DA, Brar I, Stephens JL, Girard PM, Huhn G, Plummer A, Liu YP, Cheng AK, McCallister S; GS-US-292-0109 team. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide in antiretroviral regimens for virologically suppressed adults with HIV-1 infection: a randomised, active-controlled, multicentre, open-label, phase 3, non-inferiority study. Lancet Infect Dis. 2016 Jan;16(1):43-52. doi: 10.1016/S1473-3099(15)00348-5. Epub 2015 Nov 2. PMID 26538525
- [Background] Pozniak A, Arribas JR, Gathe J, Gupta SK, Post FA, Bloch M, Avihingsanon A, Crofoot G, Benson P, Lichtenstein K, Ramgopal M, Chetchotisakd P, Custodio JM, Abram ME, Wei X, Cheng A, McCallister S, SenGupta D, Fordyce MW; GS-US-292-0112 Study Team. Switching to Tenofovir Alafenamide, Coformulated With Elvitegravir, Cobicistat, and Emtricitabine, in HIV-Infected Patients With Renal Impairment: 48-Week Results From a Single-Arm, Multicenter, Open-Label Phase 3 Study. J Acquir Immune Defic Syndr. 2016 Apr 15;71(5):530-7. doi: 10.1097/QAI.0000000000000908. PMID 26627107
- [Background] Hill A, Hughes SL, Gotham D, Pozniak AL. Tenofovir alafenamide versus tenofovir disoproxil fumarate: is there a true difference in efficacy and safety? J Virus Erad. 2018 Apr 1;4(2):72-79. doi: 10.1016/S2055-6640(20)30248-X. PMID 29682298
- [Background] Sax PE, Zolopa A, Brar I, Elion R, Ortiz R, Post F, Wang H, Callebaut C, Martin H, Fordyce MW, McCallister S. Tenofovir alafenamide vs. tenofovir disoproxil fumarate in single tablet regimens for initial HIV-1 therapy: a randomized phase 2 study. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):52-8. doi: 10.1097/QAI.0000000000000225. PMID 24872136
- [Background] Mills A, Crofoot G Jr, McDonald C, Shalit P, Flamm JA, Gathe J Jr, Scribner A, Shamblaw D, Saag M, Cao H, Martin H, Das M, Thomas A, Liu HC, Yan M, Callebaut C, Custodio J, Cheng A, McCallister S. Tenofovir Alafenamide Versus Tenofovir Disoproxil Fumarate in the First Protease Inhibitor-Based Single-Tablet Regimen for Initial HIV-1 Therapy: A Randomized Phase 2 Study. J Acquir Immune Defic Syndr. 2015 Aug 1;69(4):439-45. doi: 10.1097/QAI.0000000000000618. PMID 25867913
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016